CLINICAL TRIAL: NCT02639247
Title: A Phase 3, Global, Multicenter, Randomized, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir/Velpatasvir/GS-9857 Fixed-Dose Combination for 12 Weeks and Sofosbuvir/Velpatasvir for 12 Weeks in Direct-Acting Antiviral-Experienced Subjects With Chronic HCV Infection Who Have Not Received an NS5A Inhibitor
Brief Title: Safety and Efficacy of SOF/VEL/VOX FDC for 12 Weeks and SOF/VEL for 12 Weeks in DAA-Experienced Adults With Chronic HCV Infection Who Have Not Received an NS5A Inhibitor
Acronym: POLARIS-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-367-1170; 2015-003167-10 (EudraCT Number)
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C Virus Infection
Keywords: Chronic
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — sofosbuvir velpatasvir voxilaprevir drug combination; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SOF/VEL/VOX (Experimental): SOF/VEL/VOX for 12 weeks
  Interventions: Drug: SOF/VEL/VOX
- SOF/VEL (Experimental): SOF/VEL for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL/VOX — 400/100/100 mg FDC tablet administered orally once daily with food
  Other Names: Vosevi®; GS-7977/GS-5816/GS-9857
  Arms: SOF/VEL/VOX
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily without regard to food
  Other Names: Epclusa®; GS-7977/GS-5816
  Arms: SOF/VEL

SUMMARY:
The primary objectives of the study are to evaluate the efficacy, safety, and tolerability of treatment with sofosbuvir/velpatasvir/voxilaprevir (Vosevi®; SOF/VEL/VOX) fixed-dose combination (FDC) for 12 weeks and of sofosbuvir/velpatasvir (Epclusa®; SOF/VEL) FDC for 12 weeks in direct-acting antiviral (DAA)-experienced adults with chronic hepatitis C virus (HCV) infection with or without cirrhosis who have not received prior treatment with a regimen containing an inhibitor of the HCV NS5A protein.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL at screening
* Chronic HCV infection (≥ 6 months)
* Treatment experienced with a direct acting antiviral medication not including a NS5A Inhibitor for HCV
* Use of protocol specified methods of contraception

Key Exclusion Criteria:

* Current or prior history of clinically significant illness that may interfere with participation in the study
* Screening ECG with clinically significant abnormalities
* Laboratory results outside of acceptable ranges at screening
* Pregnant or nursing female
* Chronic liver disease not caused by HCV
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (78):
- United States (43):
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Pasadena, California
  - Rialto, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Bastrop, Louisiana
  - Baltimore, Maryland
  - Catonsville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - New York, New York
  - Asheville, North Carolina
  - Fayetteville, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (5):
  - Camperdown, New South Wales
  - Darlinghurst, New South Wales
  - Herston, Queensland
  - Clayton, Victoria
  - Melbourne, Victoria
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brampton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- France (14):
  - Clermont-Ferrand
  - Clichy
  - Grenoble
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Pessac
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (6):
  - Berlin
  - Bonn
  - Cologne
  - Frankfurt am Main
  - Hamburg
  - Hanover
- Grafton, Auckland, New Zealand
- San Juan, Puerto Rico
- United Kingdom (2):
  - London
  - Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/about/ethics-and-code-of-conduct/policies.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/about/ethics-and-code-of-conduct/policies

REFERENCES:
- [Derived] Bourliere M, Gordon SC, Flamm SL, Cooper CL, Ramji A, Tong M, Ravendhran N, Vierling JM, Tran TT, Pianko S, Bansal MB, de Ledinghen V, Hyland RH, Stamm LM, Dvory-Sobol H, Svarovskaia E, Zhang J, Huang KC, Subramanian GM, Brainard DM, McHutchison JG, Verna EC, Buggisch P, Landis CS, Younes ZH, Curry MP, Strasser SI, Schiff ER, Reddy KR, Manns MP, Kowdley KV, Zeuzem S; POLARIS-1 and POLARIS-4 Investigators. Sofosbuvir, Velpatasvir, and Voxilaprevir for Previously Treated HCV Infection. N Engl J Med. 2017 Jun 1;376(22):2134-2146. doi: 10.1056/NEJMoa1613512. PMID 28564569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across 101 study sites in North America, Europe, and Asia Pacific. The first participant was screened on 23 December 2015. The last study visit occurred on 18 January 2017.
Pre-assignment Details: 397 participants were screened.
Groups:
- SOF/VEL/VOX 12 Weeks: Sofosbuvir/veltapasvir/voxilaprevir (Vosevi®; SOF/VEL/VOX) (400/100/100 mg) fixed-dose combination (FDC) tablet orally once daily with food for 12 weeks
- SOF/VEL 12 Weeks: Sofosbuvir/Velpatasvir (Epclusa®; SOF/VEL) (400/100 mg) FDC tablet orally once daily without regard to food for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks
Started | 182 | 151
Completed | 177 | 149
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 2 | 0
Not completed — Withdrew Consent | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all randomized or enrolled participants who received at least 1 dose of study drug
Groups:
- SOF/VEL/VOX 12 Weeks: SOF/VEL/VOX (400/100/100 mg) FDC tablet orally once daily with food for 12 weeks
- SOF/VEL 12 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily without regard to food for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks | Total
Number analyzed (Participants) | 182 | 151 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.0) | 57 (7.3) | 57 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 143 | 114 | 257
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 160 | 131 | 291
  Black or African American | 16 | 13 | 29
  Asian | 2 | 4 | 6
  Other | 2 | 1 | 3
  American Indian or Alaska Native | 2 | 0 | 2
  Native Hawaiian or Pacific Islander | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 8 | 27
  Not Hispanic or Latino | 163 | 143 | 306
Region of Enrollment [Number; unit: participants]
  United States | 101 | 87 | 188
  Australia | 13 | 10 | 23
  Canada | 18 | 20 | 38
  France | 26 | 19 | 45
  Germany | 14 | 10 | 24
  New Zealand | 1 | 2 | 3
  United Kingdom | 9 | 3 | 12
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene
  Participants
    CC | 33 | 29 | 62
    CT | 107 | 95 | 202
    TT | 42 | 27 | 69
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.56) | 6.3 (0.66) | 6.3 (0.61)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 46 | 38 | 84
  ≥ 800,000 IU/mL | 136 | 113 | 249

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all randomized or enrolled participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 182 | 151
percentage of participants | 97.8 [94.5 to 99.4] | 90.1 [84.1 to 94.3]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinue Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 182 | 151
percentage of participants | 0 | 0.7

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participcants
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 182 | 151
percentage of participcants
  SVR4 | 98.4 [95.3 to 99.7] | 91.4 [85.7 to 95.3]
  SVR24 | 97.8 [94.5 to 99.4] | 90.1 [84.1 to 94.3]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On Treatment
Time Frame: Weeks 1, 2, 4, 8 and 12
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 182 | 151
percentage of participants
  Week 1 | 15.9 [10.9 to 22.1] | 17.2 [11.6 to 24.2]
  Week 2 | 62.6 [55.2 to 69.7] | 56.3 [48.0 to 64.3]
  Week 4 | 88.5 [82.9 to 92.7] | 90.7 [84.9 to 94.8]
  Week 8 | 100.0 [98.0 to 100.0] | 98.7 [95.3 to 99.8]
  Week 12 | 98.9 [96.1 to 99.9] | 99.3 [96.3 to 100.0]

5. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 182 | 151
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 181 | 148
  Change at Week 1 | -4.29 (0.627) | -4.17 (0.651)
  Change at Week 2: number analyzed (Participants) | 180 | 151
  Change at Week 2 | -4.93 (0.604) | -4.78 (0.677)
  Change at Week 4 | -5.13 (0.561) | -5.06 (0.660)
  Change at Week 8: number analyzed (Participants) | 182 | 150
  Change at Week 8 | -5.17 (0.562) | -5.08 (0.759)
  Change at Week 12: number analyzed (Participants) | 180 | 150
  Change at Week 12 | -5.17 (0.559) | -5.09 (0.727)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 182 | 151
percentage of participants | 0.5 | 9.9

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set: all participants who received at least 1 dose of study drug
Arm/Group | SOF/VEL/VOX 12 Weeks | SOF/VEL 12 Weeks
Serious Adverse Events (participants affected / at risk) | 4/182 | 4/151
Other Adverse Events (participants affected / at risk) | 111/182 | 88/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX 12 Weeks (N=182) | SOF/VEL 12 Weeks (N=151)
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX 12 Weeks (N=182) | SOF/VEL 12 Weeks (N=151)
Abdominal pain (Gastrointestinal disorders) | 3 | 9
Diarrhoea (Gastrointestinal disorders) | 36 | 7
Nausea (Gastrointestinal disorders) | 22 | 12
Asthenia (General disorders) | 10 | 9
Fatigue (General disorders) | 43 | 43
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Headache (Nervous system disorders) | 50 | 43
Insomnia (Psychiatric disorders) | 12 | 3
Irritability (Psychiatric disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years